CLINICAL TRIAL: NCT04075890
Title: Arbitration Between Habitual and Goal-directed Behavior in Obsessive-compulsive Disorder: Circuit Dynamics and Effects of Noninvasive Neurostimulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Reza Tadayon-Nejad, MD, PhD, Assistant Clinical Professor of Psychiatry, University of California, Los Angeles
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 17-001360
Record Dates: First submitted 2019-08-29; First posted 2019-09-03 (Actual); Results first posted 2025-12-12 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-11

CONDITIONS: OCD; Decision-Making; tDCS; fMRI
MeSH Terms: interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Healthy subjects (Active Comparator)
  Interventions: Device: transcranial Direct Current Stimulation (tDCS)
- OCD subjects (Active Comparator)
  Interventions: Device: transcranial Direct Current Stimulation (tDCS)

INTERVENTIONS:
Device: transcranial Direct Current Stimulation (tDCS) — tDCS is a non-invasive brain stimulation method by which constant low direct current can be delivered to the sculpt for changing the excitability of neuronal structure adjunct to the stimulating electrode.

SUMMARY:
People utilize two behavioral strategies, goal-directed and habitual, when engaging in value-based decision-making that involves rewarding or punishing outcomes. Accumulating evidence suggests an imbalance between habitual and goal-directed behavior in favor of habitual control in parallel with exaggerated tendency toward compulsive/harm avoidance behavior in OCD. In healthy subjects, an arbitration mechanism has been proposed recently that controls the balance between those two strategies of action selection. Arbitration regions regulate the goal-directed/habitual decision-making balance by selectively downregulating the activity of the habitual regions. This project aims to explore the neurobehavioral characteristics of arbitration mechanism and its relationship with behaviors and clinical phenotypes in OCD by applying computational cognitive neuroscience, clinical task-based functional magnetic resonance imaging (fMRI) and transcranial direct current stimulation (tDCS) method.

DETAILED DESCRIPTION:
Investigators will recruit 30 male and female adults (age 18-65) with OCD and 30 age-, sex-, and education-matched healthy (medically, neurologically and psychiatrically) controls for this project. Each participant will come for three sessions. There will be 3-4 days interval between sessions:

Session 1 that includes initial clinical assessment and obtaining T1 structural image (needed for neuronavigation analysis and electric field modeling).

Session 2 and 3 that include performing two separate decision-making and symptom provocation-avoidance tasks by participants with OCD and healthy controls under two conditions: while scanned inside the MRI scanner (no tDCS) or while receiving neuronavigated tDCS neurostimulation outside the scanner (no fMRI imaging). As participates will perform each task twice, there might be an order effect on task performance. For minimizing the impact of such a potential order effect on imaging and tDCS results, participants will be randomly assigned to undergo scanning in the session 2 and then receive tDCS in the session 3 or in the opposite order (tDCS in session 2 and then imaging in session 3) but in each session only one of imaging or tDCS experiments (for both tasks) will be conducted for each participant. OCD-relevant and aversive picture rating (explained below) will be done always in the session 3 as the last experiment.

ELIGIBILITY:
A) OCD participants inclusion criteria:

1. DSM-5 diagnostic criteria for OCD as primary (most severe) diagnosis (based on the Mini International Neuropsychiatric Interview).
2. Yale-Brown Obsessive-Compulsive Scale (YBOCS) total score is equal or greater than 16.
3. unmediated or being on a stable dose of medication (only SSRIs and clomipramine) for at least 12 weeks prior to the study.
4. fluent English speaker.
5. signed informed consent.

B) OCD participants exclusion criteria:

1. IQ greater than 80 on the Wechsler Abbreviated Scales of Intelligence.
2. lifetime DSM-5 diagnosis of mania, psychotic disorder, or substance dependence (per MINI).
3. current DSM-5 diagnosis of MDD if Montgomery-Asberg Depression Scale (MADRS) scores are equal or greater than 35 (severe), or ADHD.
4. taking any psychotropic medication other than SSRIs or clomipramine.
5. severe psychiatric symptom that requires immediate inpatient psychiatric intervention such as suicidality.
6. presence of any serious psychiatric, psychosocial, or neurological condition requiring immediate treatment.

C) Healthy control inclusion criteria:

1-males and females age 18-65 years with signed informed consent and IQ greater than 80 on WASI.

D) Exclusion criteria for all participants:

1. presence of any MR scan contraindications particularly body metal or positive pregnancy test.
2. medical conditions in which cerebral metabolism might be compromised such as thyroid disorders, diabetes or current tobacco smoking (potential effect on imaging endpoints).
3. any history of seizure disorders.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2019-07-15 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-01-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- UCLA, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Healthy Subjects: fMRI Imaging First, Then tDCS: Healthy control subjects who first underwent imaging experiments in which they performed tasks in the MRI scanner on their second visit (no brain stimulation) and on the third session, performed the same tasks when receiving brain stimulation by tDCS (no imaging).
- Healthy Subjects:tDCS First, Then fMRI Imaging: Healthy control subjects that first performed the two tasks when receiving brain stimulation by tDCS (no imaging) on their second visit and on the third session performed the same tasks in the MRI scanner (no brain stimulation).
- OCD Subjects: fMRI Imaging First, Then tDCS: OCD subjects who first underwent imaging experiments in which they performed tasks in the MRI scanner on their second visit (no brain stimulation) and on the third session, performed the same tasks when receiving brain stimulation by tDCS (no imaging).
- OCDSubjects: tDCS First, Then fMRI Imaging: OCD control subjects that first performed the two tasks when receiving brain stimulation by tDCS (no imaging) on their second visit and on the third session performed the same tasks in the MRI scanner (no brain stimulation).
Period: First Intervention (4 Days)
Arm/Group | Healthy Subjects: fMRI Imaging First, Then tDCS | Healthy Subjects:tDCS First, Then fMRI Imaging | OCD Subjects: fMRI Imaging First, Then tDCS | OCDSubjects: tDCS First, Then fMRI Imaging
Started | 16 | 16 | 16 | 18
Completed | 15 | 15 | 15 | 15
Not Completed | 1 | 1 | 1 | 3
Period: Second Intervention (4 Days)
Arm/Group | Healthy Subjects: fMRI Imaging First, Then tDCS | Healthy Subjects:tDCS First, Then fMRI Imaging | OCD Subjects: fMRI Imaging First, Then tDCS | OCDSubjects: tDCS First, Then fMRI Imaging
Started | 16 | 16 | 16 | 18
Completed | 15 | 15 | 15 | 15
Not Completed | 1 | 1 | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Healthy Subjects: fMRI Imaging First, Then tDCS: Healthy control subjects who first underwent imaging experiments in which they performed tasks in the MRI scanner on their second visit (no brain stimulation) and on the third session, performed the same tasks when receiving brain stimulation by tDCS (no imaging).
  A) Healthy control inclusion criteria:
  1-Males and females age 18-65 years fluent English speaker with signed informed consent.
  B) Exclusion criteria for control participants:
  1. presence of any MR scan contraindications particularly body metal or positive pregnancy test.
  2. medical conditions in which cerebral metabolism might be compromised such as thyroid disorders, diabetes or current tobacco smoking (potential effect on imaging endpoints).
  3. any history of seizure disorders.
- Healthy Subjects: tDCS First, Then fMRI Imaging: Healthy control subjects that first performed the two tasks when receiving brain stimulation by tDCS (no imaging) on their second visit and on the third session performed the same tasks in the MRI scanner (no brain stimulation).
  A) Healthy control inclusion criteria:
  1-Males and females age 18-65 years fluent English speaker with signed informed consent.
  B) Exclusion criteria for control participants:
  1. presence of any MR scan contraindications particularly body metal or positive pregnancy test.
  2. medical conditions in which cerebral metabolism might be compromised such as thyroid disorders, diabetes or current tobacco smoking (potential effect on imaging endpoints).
  3. any history of seizure disorders.
- OCD Subjects: fMRI Imaging First, Then tDCS: OCD subjects who first underwent imaging experiments in which they performed tasks in the MRI scanner on their second visit (no brain stimulation) and on the third session, performed the same tasks when receiving brain stimulation by tDCS (no imaging).
  A) OCD participants inclusion criteria:
  1. DSM-5 diagnostic criteria for OCD as primary (most severe) diagnosis (based on the Mini International Neuropsychiatric Interview).
  2. Yale-Brown Obsessive-Compulsive Scale (YBOCS) total score is equal or greater than 16.
  3. unmediated or being on a stable dose of medication (only SSRIs and clomipramine) for at least 12 weeks prior to the study.
  4. fluent English speaker.
  5. signed informed consent.
  B) OCD participants exclusion criteria:
  1. IQ greater than 80 on the Wechsler Abbreviated Scales of Intelligence.
  2. lifetime DSM-5 diagnosis of mania, psychotic disorder, or substance dependence (per MINI).
  3. current DSM-5 diagnosis of MDD if Montgomery-Asberg Depression Scale (MADRS) scores are equal or greater than 35 (severe), or ADHD.
  4. taking any psychotropic medication other than SSRIs or clomipramine.
  5. severe psychiatric symptom that requires immediate inpatient psychiatric intervention such as suicidality.
  6. presence of any serious psychiatric, psychosocial, or neurological condition requiring immediate treatment.
  C) Exclusion criteria for OCD participants:
  1. presence of any MR scan contraindications particularly body metal or positive pregnancy test.
  2. medical conditions in which ce
- OCD Subjects: tDCS First, Then fMRI Imaging: OCD control subjects that first performed the two tasks when receiving brain stimulation by tDCS (no imaging) on their second visit and on the third session performed the same tasks in the MRI scanner (no brain stimulation).
  A) OCD participants inclusion criteria:
  1. DSM-5 diagnostic criteria for OCD as primary (most severe) diagnosis (based on the Mini International Neuropsychiatric Interview).
  2. Yale-Brown Obsessive-Compulsive Scale (YBOCS) total score is equal or greater than 16.
  3. unmediated or being on a stable dose of medication (only SSRIs and clomipramine) for at least 12 weeks prior to the study.
  4. fluent English speaker.
  5. signed informed consent.
  B) OCD participants exclusion criteria:
  1. IQ greater than 80 on the Wechsler Abbreviated Scales of Intelligence.
  2. lifetime DSM-5 diagnosis of mania, psychotic disorder, or substance dependence (per MINI).
  3. current DSM-5 diagnosis of MDD if Montgomery-Asberg Depression Scale (MADRS) scores are equal or greater than 35 (severe), or ADHD.
  4. taking any psychotropic medication other than SSRIs or clomipramine.
  5. severe psychiatric symptom that requires immediate inpatient psychiatric intervention such as suicidality.
  6. presence of any serious psychiatric, psychosocial, or neurological condition requiring immediate treatment.
  C) Exclusion criteria for OCD participants:
  1. presence of any MR scan contraindications particularly body metal or positive pregnancy test.
  2. medical conditions in which cerebral metabolism might be c
- Total: Total of all reporting groups
Arm/Group | Healthy Subjects: fMRI Imaging First, Then tDCS | Healthy Subjects: tDCS First, Then fMRI Imaging | OCD Subjects: fMRI Imaging First, Then tDCS | OCD Subjects: tDCS First, Then fMRI Imaging | Total
Number analyzed (Participants) | 15 | 15 | 15 | 15 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 15 | 15 | 15 | 15 | 60
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: year] | 25 [18 to 65] | 27 [18 to 65] | 27 [18 to 65] | 29 [18 to 65] | 27 [18 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 9 | 8 | 8 | 35
  Male | 5 | 6 | 7 | 7 | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 2 | 4 | 3 | 12
  Not Hispanic or Latino | 11 | 13 | 11 | 12 | 47
  Unknown or Not Reported | 1 | 0 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 5 | 4 | 3 | 4 | 16
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 0 | 1 | 0 | 3
  White | 7 | 11 | 11 | 11 | 40
  More than one race | 1 | 0 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 15 | 15 | 15 | 15 | 60

OUTCOME MEASURES:

1. Primary Outcome: Strength of Behaving Model-based (Goal-directed)
Description: Strength of behaving model-based (goal-directed) is measured and quantifiedas a continuous real number between 0 and 1. Here, having a strength's valueof 1 of behaving model-based means that subject in her/his decision-making,exclusively and always utilizes a model-based (goal-directed) strategy fordecision making and having a value of Zero means not utilizing model-based(goal-directed) strategy at all when decising.
Time Frame: On the second or third session when subjects performed the task in the MRI scanner.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Healthy Subjects: fMRI Imaging First, Then tDCS | Healthy Subjects: tDCS First, Then fMRI Imaging | OCD Subjects: fMRI Imaging First, Then tDCS | OCD Subjects: tDCS First, Then fMRI Imaging
Number analyzed (Participants) | 15 | 15 | 15 | 15
units on a scale | 0.09 (0.132) | 0.07 (0.14) | -0.08 (0.082) | 0.06 (0.091)

2. Primary Outcome: Reaction Time in Response to Stimuli With OCD Themes
Description: This is a time interval (in seconds) between the start of presentation of visual stimuli with OCD themes and when subjects pushed a bottom to stop the presentation when they could not tolerate those more during symptom provocation and avoidance task.
Time Frame: On the second or third session when subjects performed the task in the MRI scanner.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Healthy Subjects: fMRI Imaging First, Then tDCS | Healthy Subjects: tDCS First, Then fMRI Imaging | OCD Subjects: fMRI Imaging First, Then tDCS | OCD Subjects: tDCS First, Then fMRI Imaging
Number analyzed (Participants) | 15 | 15 | 15 | 15
seconds | 5.6 (2.18) | 5.5 (2.91) | 4.3 (2.01) | 4.8 (2.93)

3. Primary Outcome: Strength of Frontal Arbitration Modulation of Basal Ganglia Habit Region.
Description: Here, by applying Dynamic Causal Modeling (DCM) method, we measured thestrength of frontal arbitration (the interior frontal gyrus (IFG)) modulation ofbasal ganglia habit region (the posterolateral putamen) in terms of the effective(directed) connectivity between the interior frontal gyrus (IFG) andposterolateral putamen. This DCM-based effective connectivity can have avalue between -1 and +1. A value of -1 means a maximum effective connectivitybetween the interior frontal gyrus (IFG) and posterolateral putamen. A value of+1 means maximum excitatory effective connectivity between the interior frontalgyrus (IFG) and posterolateral putamen. And a value of 0 means no effectiveconnectivity between the interior frontal gyrus (IFG) and posterolateralputamen.
Time Frame: On the second or third session when subjects performed the task in the MRI scanner
Measure: Mean (Standard Deviation); unit: units on ascale
Arm/Group | Healthy Subjects: fMRI Imaging First, Then tDCS | Healthy Subjects: tDCS First, Then fMRI Imaging | OCD Subjects: fMRI Imaging First, Then tDCS | OCD Subjects: tDCS First, Then fMRI Imaging
Number analyzed (Participants) | 15 | 15 | 15 | 15
units on ascale | -0.07 (0.121) | -0.06 (0.131) | -0.003 (0.161) | -0.004 (0.132)

ADVERSE EVENTS:
Time Frame: 4 years and six months.
Groups:
- Healthy Subjects: fMR Imaging; OCD Subjects: fMRI Imaging: This was during the sessions when subjects performed tasks in MRI scanner.
- Healthy Subjects: tDCS; OCD Subjects:tDCS: This was during the sessions when subjects performed tasks with brain stimulation (tDCS).
Arm/Group | Healthy Subjects: fMR Imaging | Healthy Subjects: tDCS | OCD Subjects: fMRI Imaging | OCD Subjects:tDCS
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30 | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30 | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30 | 0/30 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-09-20): https://cdn.clinicaltrials.gov/large-docs/90/NCT04075890/Prot_SAP_001.pdf